CLINICAL TRIAL: NCT07344545
Title: Identification of Gut Microbiota Signatures Associated With Health Metrics in a Community-based Adult Cohort: a Cross-sectional Study
Brief Title: Mining the Gut Microbiota of Adults for Health-relevant Microbial Signatures.
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Huzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong He, Department of Laboratory Medicine, Zhujiang Hospital
Other Study IDs: Zhujiang-Huzhou
Record Dates: First submitted 2025-12-03; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult volunteers: The study population consists of 1,530 middle-aged and elderly volunteers from the same community who underwent comprehensive health examinations at Huzhou Central Hospital . All participants completed a multi-dimensional assessment including biospecimen collection, physical/imaging examinations, and psychometric evaluations.
  Interventions: Other: Observational, non-interventional study.

INTERVENTIONS:
Other: Observational, non-interventional study. — Observational, non-interventional study.

SUMMARY:
Mining the gut microbiota of adults for health-relevant microbial signatures.

DETAILED DESCRIPTION:
This study is a community-based, observational cross-sectional investigation, enrolling 1,530 middle-aged and elderly volunteers.

Data were collected through a systematic, multi-dimensional assessment, which included:

Biospecimen Collection: Blood, urine, and stool samples were obtained from the volunteers.

Physical and Imaging Examinations: Procedures included anthropometric measurements, vital sign monitoring, oral examinations, electrocardiograms, physical examinations of key organs, and abdominal ultrasonography.

Psychological and Cognitive Assessments: Standardized scales were administered to assess anxiety/depression and memory function.

All clinical and questionnaire data were processed through standardized procedures, forming a comprehensive health database for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria：

* Community-dwelling adults aged 30 to 95 years.
* Individuals who underwent an annual health examination at the Health Management Center of Huzhou Central Hospital during the specified time period.
* Ability to comprehend the study content and voluntarily provide signed informed consent.
* Willingness and ability to provide the required biospecimens (blood, urine, stool).

Exclusion Criteria:

* Concurrent participation in another interventional clinical trial that is likely to interfere with the results of this study.
* Voluntary withdrawal from the study.

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 1530 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Identification of Health-Relevant Signatures in Adults | Baseline
  Primary Outcome Measure 1)Change in standard laboratory parameters from baseline:Changes in routine laboratory parameters measured in blood, urine, and stool samples, including complete blood count and standard serum biochemistry panels.Unit of Measure: Various laboratory units (e.g., g/L, U/L, mmol/L); 2) Change in anthropometric measurements from baseline: Anthropometric measurements including body weight (kg), height (m), and body mass index (BMI, kg/m²).Unit of Measure:kg, m, kg/m²; 3) Alcohol consumption status: Alcohol consumption status assessed by self- report, categorized as current drinker or non-drinker at enrollment.Unit of Measure:Categorical (yes/no); 4) Hospital Anxiety and Depression Scale (HADS) scores: Anxiety and depression symptom severity assessed using the Hospital Anxiety and Depression Scale, including anxiety and depression subscale scores.Unit of Measure:Score on a standardized scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China